CLINICAL TRIAL: NCT01348412
Title: Phase II Randomized Study Comparing the Association of Intraarterial Perfusion of Raltitrexed and Oxaliplatin Versus Standard Chemotherapy Using Intravenous Perfusion for Colorectal Cancer Patient With Metastases Localized to Liver After Failure of Conventional Treatments.
Brief Title: Hepatic Arterial Chemotherapy With Raltitrexed and Oxaliplatin Versus Standard Chemotherapy in Unresectable Liver Metastases From Colorectal Cancer After Conventional Chemotherapy Failure
Acronym: HEARTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: National Cancer Institute, France (Other Government); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0329-1ghfr09
Record Dates: First submitted 2011-04-27; First posted 2011-05-05 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: non resectable metastases; liver of colic or rectal origin; after failure of the conventional treatments
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Experimental): Hepatic artery infusion through an implanted arterial catheter of the combination of raltitrexed (3 mg/m ²) and oxaliplatin (100 mg/m ²) every 21 days.
  Interventions: Drug: oxaliplatin; Drug: raltitrexed
- ARM B (Active Comparator): Intravenous standard chemotherapy.
  Interventions: Drug: other intravenous chemotherapy drugs

INTERVENTIONS:
Drug: oxaliplatin — 130 mg/m²Every 21 days
  Arms: ARM A
Drug: raltitrexed — 3 mg/m² with a maximum of 6 mg every 21 days
  Arms: ARM A
Drug: other intravenous chemotherapy drugs
  Arms: ARM B

SUMMARY:
Standard treatment of metastatic colorectal cancers relies on fluoropyrimidines, irinotecan alone or in association with fluoropyrimidines, oxaliplatin in association with fluoropyrimidines, bevacizumab and anti EGFR antibodies. After failure of classical regimen the national reference frame on the basis of phase II study proposes an association of fluoropyrimidine and mitomycin. These treatments give response rates of 10-20% with progression free survivals from 2 to 3 months. Hepatic intra-arterial chemotherapy is logical in the case of isolated hepatic metastases nonaccessible to curative resection: 1) hepatic metastases are vascularized by hepatic arterial system in contrast to nontumoral hepatic parenchyma; 2) arterial perfusion of oxaliplatin leads to a strong extraction by the liver during the first passage, a high intra-tumoral concentration and a low systemic concentration. So oxaliplatin is a drug of choice for arterial treatment but combination with fluoropyrimidines is impossible because of need for prolonged perfusion. Floxuridin is not available in France. Raltitrexed, a definitive inhibitor of the thymidylate synthase, does not require a prolonged perfusion and could be a good substitute.In a previous pilot study we demonstrated the feasibility, safety and efficacy of combination of raltitrexed and oxaliplatin arterial perfusion. Now we propose a phase II randomized clinical trial to evaluate the efficacy of hepatic arterial infusion of raltitrexed and oxaliplatin association versus standard chemotherapy for patients with metastases of colorectal origin restricted to the liver after failure of conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature by the patient-
* Cover by an health insurance
* Age between 18 and 75 years
* Age between 76 et 80 years if patient WHO Status 0
* WHO status of 0 or 1
* Estimated Life expectancy > 3 months
* Hepatic metastases of colorectal cancer confirmed on CT Scan without extra-hepatic metastasis (the presence of asymptomatic primary tumor is tolerated)
* TEP-Scan without fixation outside the liver and the primary tumor
* Histological proven colorectal cancer obtained from primary tumor or the hepatic metastases
* Metastases not accessible to curative hepatectomy (impossible R0 surgery or leaving less than 30 % of residual liver), or requiring a complex, very wide hepatectomy (5 segments or more) and\or risky procedure (RPC Class II)- - Presence of hepatic lesion > 10 mm on CTScan or hepatic MRI
* Failure or arrest of a previous chemotherapy because of intolerance to oxaliplatin, irinotecan, a fluoropyrimidine and/or target therapies (bevacizumab, cetuximab or panitumumab given for tumor expressing wild type Ki-Ras)
* Bilirubinemia< 1,5 times the superior limit of the normal ( N ),
* ASAT and ALAT < 5 N,
* Creatinemia < 1.5 N and creatinine clearance > 65ml/mn,
* Neutrophils > 1,5 x 109/L, platelets 100 x 109/L, hemoglobin > 9 g/dL (patients includables even after red blood cell transfusion)-Reference CTScan +/-MRI performed in 21 days preceding the first cycle of treatment

Exclusion Criteria:

* extra-hepatic metastases (presence of 1 to 3 pulmonary nodules, of a maximal diameter of 5 mm with non specific aspect on CTScan and with no fixation on TEP Scan does not constitute a criterion of exclusion)
* Symptomatic primary colorectal tumor in place
* Contraindication for allergy of rank 3-4 for one of the compounds of chemotherapy- Peripheral neuropathy > 2 (Levy Scale)
* Current participation or in the 30 days preceding the inclusion in the study in another therapeutic trial with an experimental molecule
* Concomitant systemic treatment by immunotherapy, chemotherapy or hormonotherapy- Unbalanced serious illness, unchecked active infection or the other underlying serious disorder susceptible to prevent the patient from receiving the treatment
* Pregnancy (pregnancy test compulsory for the inclusion), breast-feeding
* Intestinal occlusion or sub-occlusion or history of inflammatory intestinal disease
* Other cancer during the 5 years preceding entry in the trial or concomitant (except in situ cancer of the cervix or skin basal cell carcinoma)Patient in custody or under guardianship, Impossibility to adhere to the medical follow-up for geographical, social or psychiatric reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-12-15 (Actual); Primary Completion 2010-12-15 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
progression-free survival | for each patient after the 6 months of treatment

SECONDARY OUTCOMES:
Estimate the parameters of tumor perfusion using arterial CT Scan data | for each patient of experimental arm every 9 weeks after the six months of treatment or until progression
Estimate the rate of objective response according to the criteria of CHOI and RECIST | for each patient every 9 weeks during the 6 months of treatment or until progression
Estimate the overall survival which will be compared with the median of overall survival in other studies published in the literature | after all data completion after the end of all patient follow-up (december 2013-anticipated)
Estimate the rate of secondary resectable hepatic metastases | after all data completion after the end of all patient follow-up (december 2013-anticipated)
Estimate the tolerance of the treatment (NCI-CTCAE version 4.0) | For each patient every 21 days during the six months of treatment and for one year of follow up or until progression
Estimate the quality of life (QLQ C30) and the fatigue MFI20 | after all data completion after the end of all patient follow-up (december 2013-anticipated)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France